CLINICAL TRIAL: NCT04633603
Title: LázBarát™ (FeverFriend™) Projekt: Attitude Toward Fever and Its Change in the Healthcare System
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pecs (Other)
Collaborators: Dr. Szőke Henrik és Társa Egészségügyi Szolgáltató Kft. (Unknown); Hungarian Medical Chamber / Magyar Orvosi Kamara (Győr-Moson-Sopron Megye) (Unknown); University of Witten (Unknown); Heim Pál Children's Hospital / Heim Pál Országos Gyermekgyógyászati Intézet (Unknown); Hungarian Emergency Service / Országos Mentőszolgálat (Unknown); Civil Support Közhasznú Nonprofit Kft. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IV/209-1/2020/EKU
Record Dates: First submitted 2020-10-29; First posted 2020-11-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Fever; Anxiety; Help-Seeking Behavior; Virus Diseases; Bacterial Infections; Overdose of Analgesic Drug
Keywords: childhood fever; help-seeking behavior; fever phobia; mobile application; guideline adherence; antipyretics; antibiotics; health literacy; socio-economic assessment
MeSH Terms: conditions — Fever; Anxiety Disorders; Help-Seeking Behavior; Virus Diseases; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients: There is no pre-specified group or subgroup of participant(s) assigned to receive the specific intervention(s) (or no intervention) according to the protocol. All patients get the same possibility to register their data and follow management advice.
  Interventions: Device: FeverFriend mobile application

INTERVENTIONS:
Device: FeverFriend mobile application — Registration, documentation of patients profile, documentation of fever events, following advice regarding the patient and the care-giver, documentation of follow up notifications.
  Other Names: FeverFriend web knowledge base (homepage)

SUMMARY:
The positive effects of fever are supported by a number of physiological, pathophysiological and clinical evidence. However, the negative attitude toward fever is widespread and have become persistent. According to sociological research, this is based on two main factors: comfort and fear. To change this negative attitude, awareness needs to be raised and the attitude toward fever among health care workers and the lay public needs to be reframed positively. Furthermore, the role of media users is essential, especially among the young generation.

The current Hungarian recommendation/protocol is valid since 2011 (Professional protocol of the Ministry of National Resources: Caring for a child with fever, the recommendation of the College of Pediatric and Pediatric However, the practical implementation among health professionals and the laity public is low.

Based on this protocol and current international guidelines (NICE) clinicians developed a protocol and register, where parents and caregivers can document the symptoms and runoff of fever as well as receive feedback on severity and appropriate management.

The project aims to increase the evidence-based (EBM) guideline adherence, to reduce the unnecessary use of antipyretics and antibiotics, as well as the load on the current healthcare system. The documentation of the collected data allows the investigators to map and analyze (stats) socio-demographic behavior both on individual and societal level.

DETAILED DESCRIPTION:
Goal:

Reframing the negative attitude toward fever. Reducing unnecessary use of drugs (antipyretics and antibiotics) as well as lower the number of medical consultations. In order, the investigators will use a media-based mobile application and a web knowledge base. Languages English and Hungarian.

Hypotheses:

1. The mobile application and knowledge base increases health literacy of parents and professionals.
2. The application will change the uncertain and/or negative attitude toward fever.
3. The positive change in attitude will influence antipyretic and consecutive antibiotic use, lower medical provider contact, enhancing the practical implementation of guidelines.

Method:

Noninvasive, noninterventional, self-reported, observational, prospective cohort study under real-life conditions.

Data: provided by caregivers and/or patients are grouped and classified based on the severity of the disease behind the fever.

Data analysis:

Analysis sample size calculation: To analyze guideline-adherent and non-adherent behavior at a 95% binomial confidence interval with an accuracy of +/- 2%, at least 500 fever phases are required if the smaller group comprises 5%. The investigators a-priory estimation based on surveys is that only about 15% of caretakers have a guideline-conforming approach to the management of fever, hence 1,500 fever events are needed for the planned accuracy. If adherent and non-adherent groups are approximately the same size, a maximum of ca. 2,500 fever phases are required.

The exact incidence of fever per age group is not yet known. Larger samples are required - and expected - for subgroup analyses (e.g. between age groups). Recruitment will therefore continue throughout to year 3 and beyond. The Chi² test is used to compare two subgroups. Sample size planning cannot take unplanned multiple testing into account, so the results can only be interpreted exploratively.

Subsample calculations: If a difference of 5% between two frequencies is interpreted as clinically significant, at a power of 80% and an alpha error probability of 5% assuming normal distribution in both subsamples, the following sample sizes are required: For a very rare sample, ca. 200 cases per subsample are sufficient. If the rate is around 50%, ca. 1,600 cases per subsample are required.

Software: IBM SPSS Statistics 22, Microsoft Excel ...

Research partners providing theoretical and professional background:

University of Pécs Hungarian Medical Chamber (Győr-Moson-Sopron Megye) University of Witten Heim Pál Childrens Hospital National Emergency Service Healthware Tanácsadó Kft. Dr. Szőke Henrik és Társa Egészségügyi Szolgáltató Kft.

Organizational tasks are conducted in the framework of the University of Pécs, Faculty of Health Sciences and by the Civil Support Közhasznú Nonprofit Kft.

ELIGIBILITY:
Inclusion criteria for patients: 0-100 years age, home or ambulant care, accepting the legal notice (including study-protocol, privacy- and data management), documenting patients profile. Eligibility for documentation of separate fever events: recording at least temperature and measurement method (device and place).

Exclusion criteria: severe underlying disease, patient who needs hospitalization.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are included if they downloaded and registered the mobile application. The use of the application is voluntary. A minimum of 100 individuals are included, a maximum sample size is not specified. Participants are between the age of 0-100. The target population is mainly children (0-18y).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Fever events outcome, condition of the patient 1 | During the period of single fever event (up to 5 days)
  body temperature grade Celsius
Fever events outcome, condition of the patient 2 | During the period of single fever event (up to 5 days)
  duration of fever in days
Fever events outcome, condition of the patient 3 | Before and during the period of single fever event (up to 20 days)
  medication, vaccination type and dosage
Fever events outcome, condition of the patient 4 | During the period of single fever event (up to 5 days)
  hydration: normal - somewhat decreased - severely decreased
Fever events outcome, condition of the patient 5 | During the period of single fever event (up to 5 days)
  ventilation: rate per minute
Fever events outcome, condition of the patient 6 | During the period of single fever event (up to 5 days)
  ventilation: wheezing and dyspnea (subjective scale 1-2-3-4-5; minimum 1; maximum 5; 1 is no symptom = better, 5 is the worst)
Fever events outcome, condition of the patient 7 | During the period of single fever event (up to 5 days)
  skin condition: color and rash
Fever events outcome, condition of the patient 8 | During the period of single fever event (up to 5 days)
  pulse rate beat per minute
Fever events outcome, condition of the patient 9 | During the period of single fever event (up to 5 days)
  crying quality (no, normal, abnormal)
Fever events outcome, condition of the patient 10 | During the period of single fever event (up to 5 days)
  eating last time in hours
Fever events outcome, condition of the patient 11 | During the period of single fever event (up to 5 days)
  urination painful or smelly (yes - no)
Fever events outcome, condition of the patient 12 | During the period of single fever event (up to 5 days)
  awareness: normal - sleepy - no (subjective scale; minimum = best = normal; maximum = worst = no)
Fever events outcome, condition of the patient 13 | During the period of single fever event (up to 5 days)
  exotic trip in the last 12 month yes - no
Fever events outcome, condition of the patient 14 | During the period of single fever event (up to 5 days)
  seizure yes - no
Fever events outcome, condition of the patient 15 | During the period of single fever event (up to 5 days)
  wry neck yes - no
Fever events outcome, condition of the patient 16 | During the period of single fever event (up to 5 days)
  pain yes - no pain location local - general duration hours
Care-givers state 1 | During the period of fever event (up to 5 days)
  Care-givers own feeling about the progress of patients illness (subjective scale,1 best = optimal - 2 = not sure - 3 = worst = very worried)
Care-givers state 2 | During the period of fever event (up to 5 days)
  Care-givers personal opinion about patients state: (subjective scale: minimum = best = not severe, middle = somewhat severe, maximum = worst = very severe)
Care-givers state 3 | During the period of fever event (up to 5 days)
  Care-givers self-confidence in handling the situation (subjective scale: maximum = confident; worse = somewhat confident, even worse = not really, minimum = worst = not at all)
Action taken, evaluation 1 | 48 hours after illness resolving
  Use of medication, use of medical providers service, utility of the device and knowledge base
Action taken, evaluation 2 | 48 hours after illness resolving
  Use of medication no - yes (type and dosage)
Action taken, evaluation 3 | 48 hours after last fever event documentation
  Use of medical providers service no - yes (institution type)
Action taken, evaluation 4 | 48 hours after last fever event documentation
  Utility of the device and knowledge base (subjective scale 1-2-3-4-5; minimum 1 = worst; maximum 5 = best)

OTHER OUTCOMES:
Baseline characteristics (profile of patient) 1 | at registry on the first day
  date of birth
Baseline characteristics (profile of patient) 2 | at registry on the first day
  gender: male - female - other
Baseline characteristics (profile) 3 | at registry on the first day
  height centimeter
Baseline characteristics (profile) 4 | at registry on the first day
  weight kilogram
Baseline characteristics (profile) 5 | at registry on the first day
  chronic disease yes - no
Baseline characteristics (profile) 6 | at registry on the first day
  Former use of medication in the last 12 month (antipyretics, antibiotics) yes - no, number
Baseline characteristics (profile) 7 | at registry on the first day
  Former use of healthcare providers service in the last 12 month no - yes, number of events and type of institution
Baseline characteristics (profile) 8 | at registry on the first day
  Caregivers former state at fever events of the patient in the last 12 month: care-givers state of mind, level of anxiety, behavior (subjective scale 1-2-3-4; )

CONTACTS AND LOCATIONS:
Overall Officials: Szőke Henrik, Dr, Principal Investigator — University of Pecs Faculty of Health Sciences
Locations (1):
- University of Pecs, Pécs, Hungary

REFERENCES:
- [Background] Purssell E, Collin J. Fever phobia: The impact of time and mortality--a systematic review and meta-analysis. Int J Nurs Stud. 2016 Apr;56:81-9. doi: 10.1016/j.ijnurstu.2015.11.001. Epub 2015 Nov 17. PMID 26643444
- [Background] Poirier MP, Collins EP, McGuire E. Fever phobia: a survey of caregivers of children seen in a pediatric emergency department. Clin Pediatr (Phila). 2010 Jun;49(6):530-4. doi: 10.1177/0009922809355312. Epub 2010 May 19. PMID 20488812
- [Background] Sakai R, Okumura A, Marui E, Niijima S, Shimizu T. Does fever phobia cross borders? The case of Japan. Pediatr Int. 2012 Feb;54(1):39-44. doi: 10.1111/j.1442-200X.2011.03449.x. Epub 2011 Oct 30. PMID 21883684
- [Background] Abu-Baker, N.N., Gharaibeh, H.F., Al-Zoubi, H.M., Savage, C., Gharaibeh, M.K., 2013. Mothers' knowledge and practices of managing minor illnesses of children under five years. J. Res. Nurs. 18 (7), 651-666.
- [Background] Alex-Hart, B.A., Frank-Briggs, A.I., 2011. Mothers' perception of fever management in children. Niger. Health J. 11 (2), 69-72.
- [Background] Ayatollahi, J., Behjati, M., Shahcheraghi, S.H., 2014. Mothers' knowledge, perception and management of fever in children. Paediatr. Today 1 (1), 14-17.
- [Background] Fekete Ferenc dr., Láz, ami átlépi az ingerküszöbünket, Gyermekorvos Továbbképzés, 2014. 13. évf. 1. szám
- [Background] A Nemzeti Erőforrás Minisztérium szakmai protokollja: Lázas gyermekek ellátásáról, Magyar közlöny, 2011
- [Background] Section on Clinical Pharmacology and Therapeutics; Committee on Drugs; Sullivan JE, Farrar HC. Fever and antipyretic use in children. Pediatrics. 2011 Mar;127(3):580-7. doi: 10.1542/peds.2010-3852. Epub 2011 Feb 28. PMID 21357332
- [Background] Rawson TM, Moore LS, Tivey AM, Tsao A, Gilchrist M, Charani E, Holmes AH. Behaviour change interventions to influence antimicrobial prescribing: a cross-sectional analysis of reports from UK state-of-the-art scientific conferences. Antimicrob Resist Infect Control. 2017 Jan 13;6:11. doi: 10.1186/s13756-017-0170-7. eCollection 2017. PMID 28101333
- [Background] James S, Rao SV, Granger CB. Registry-based randomized clinical trials--a new clinical trial paradigm. Nat Rev Cardiol. 2015 May;12(5):312-6. doi: 10.1038/nrcardio.2015.33. Epub 2015 Mar 17. PMID 25781411
- See also: Fever under 5s - assessment and initial management, NICE Guideline 2019 — https://www.nice.org.uk/guidance/ng143/resources/fever-in-under-5s-assessment-and-initial-management-pdf-66141778137541